CLINICAL TRIAL: NCT06985160
Title: Association Between Single Nucleotide Polymorphisms in TLR4, LTA and RFP175 Genes and Susceptibility to Invasive Bacterial Infections in Infants Under 3 Months of Age
Brief Title: The Association of Gene Polymorphisms With Invasive Bacterial Infections in Neonates and Young Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Caner Turan, Associate Professor, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 21975
Record Dates: First submitted 2024-04-03; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Polymorphism, Genetic; Bacterial Infections; Infant
Keywords: genetic polymorphisms, infant, invasive bacterial infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- gene polymorphisms (Other): The cohort included 100 infants aged 0-3 months diagnosed with IBIs alongside 100 control infants presenting for non-infectious conditions.
  Interventions: Other: Specific single nucleotide polymorphisms

INTERVENTIONS:
Other: Specific single nucleotide polymorphisms — Next-generation sequencing was performed to analyze the TLR4, LTA, and RFP175 genes, with a focus on specific single nucleotide polymorphisms

SUMMARY:
Invasive bacterial infections (IBIs) are globally significant, with high mortality rates, particularly within the critical 0-3 month age bracket. The first three months of life mark a peak in IBI prevalence, with an estimated 10-20% of febrile presentations in this age group resulting in an IBI diagnosis. Although multiple factors are implicated in this heightened vulnerability, the precise mechanisms driving the differential development of IBIs among similarly situated infants remain unclear. Genetic diversity and susceptibility are increasingly recognized as influential factors. Extensive literature demonstrates a correlation between genetic polymorphisms and susceptibility to invasive bacterial infections.

This study aims to explore the association of gene polymorphisms TLR4 rs2149356 (c.261-468T>G), LTA rs2229094 (c.37T>C), and RFP175 rs1585110 (c.246+8853G>A) with the occurrence of invasive bacterial infections in the population of children aged under 3 months.

We conducted a prospective observational study at a leading tertiary care hospital. The cohort included 100 infants aged 0-3 months diagnosed with IBIs alongside 100 control infants presenting for non-infectious conditions such as trauma, infantile colic, and hyperbilirubinemia. Cases with any symptoms suggesting an infection were excluded from the control group. Invasive bacterial infections categorized in this study included meningitis, pneumonia, sepsis, bacteremia, urinary tract infections, and invasive bacterial gastroenteritis. Diagnostic criteria were stringent: meningitis was confirmed via signs of bacterial infection in cerebrospinal fluid; pneumonia through auscultatory findings and radiographic evidence of pulmonary infiltrates; bacteremia by positive blood cultures; urinary tract infections by significant bacterial cultures from sterile catheterization; and gastroenteritis by the identification of pathogenic organisms in stool cultures. No additional blood was taken from the patients for the study. Instead, blood samples that were collected for tests determined by the physicians due to the patients' condition in the emergency department were retrieved from the laboratory after the requested tests were completed and reused for the study.

DETAILED DESCRIPTION:
We conducted a prospective observational study at a leading tertiary care hospital in Turkey. The cohort included 100 infants aged 0-3 months diagnosed with IBIs alongside 100 control infants presenting for non-infectious conditions. Ethical approval was secured from the institutional review board in compliance with the Declaration of Helsinki. Informed consent was obtained in written form from the parents or legal guardians of all participants prior to enrollment.

Invasive bacterial infections categorized in this study included meningitis, pneumonia, sepsis, bacteremia, urinary tract infections, and invasive bacterial gastroenteritis. Diagnostic criteria were stringent: meningitis was confirmed via signs of bacterial infection in cerebrospinal fluid; pneumonia through auscultatory findings and radiographic evidence of pulmonary infiltrates; bacteremia by positive blood cultures; urinary tract infections by significant bacterial cultures from sterile catheterization; and gastroenteritis by the identification of pathogenic organisms in stool cultures.

DNA was extracted from whole blood samples using the QIAamp DNA Mini Kit (Qiagen), according to the manufacturer's instructions. The purity and concentration of the DNA were quantified using a NanoDrop ND-1000 Spectrophotometer. Only DNA samples that met the quality and concentration criteria proceeded to sequencing. The sequence analysis targeted specific regions pertinent to the polymorphisms identified in the study's objectives.

DNA samples were processed using a sequence of analytical techniques to identify the polymorphisms TLR4 rs2149356 (c.261-468T>G), LTA rs2229094 (c.37T>C), and RFP175 rs1585110 (c.246+8853G>A), as detailed in our previous work [18]:

Primers targeting the regions encompassing TLR4 rs2149356 (c.261-468T>G), LTA rs2229094 (c.37T>C), and RFP175 rs1585110 (c.246+8853G>A) were designed using the Primer3 web tool. Criteria for primer design included a length of 18-24 base pairs, GC content between 30-50%, specificity to the target DNA region, and a melting temperature (Tm) ranging from 58-62 °C to ensure optimal amplification of a 300-500 base pair region.

Polymerase Chain Reaction (PCR) was employed for the amplification of the target regions. Each reaction mixture, prepared in a 25 µl volume, contained 0.4 µM of each primer, 2 ng of genomic DNA, 4 mM MgCl2, 0.05 µl Taq DNA polymerase, and 0.4 mM of each dNTP. Twelve such mixtures were assembled in PCR tubes. Amplification was performed under optimized conditions in a thermal cycler.

Post-amplification, the PCR products were subjected to agarose gel electrophoresis for verification. A 2% agarose gel was prepared by dissolving agarose in TBE buffer, followed by addition of ethidium bromide post-cooling. For electrophoresis, PCR products were mixed with loading dye and introduced into the gel alongside a DNA ladder. The electrophoresis was run at 120 volts, after which the gel was visualized under UV light using a gel documentation system.

After verification of the target amplicons by agarose gel electrophoresis, the PCR products were prepared for sequencing. The sequencing was performed using the Illumina MiSeq platform. This high-throughput sequencing process generated FastQ files, which were then assembled into BAM files for detailed examination. Sequence alignment and variant identification were conducted using the Integrative Genomics Viewer. Allelic variants within the sequences of the TLR4 rs2149356, LTA rs2229094, and RFP175 rs1585110 genes were meticulously identified and annotated for each subject in the study cohort.

Allelic and genotypic frequencies of the polymorphisms TLR4 rs2149356, LTA rs2229094, and RFP175 rs1585110 were assessed in patients with invasive bacterial infections compared to control subjects. Genotypic frequencies in the dominant model were evaluated by comparing the combined homozygous and heterozygous variants against the homozygous wild-type. Conversely, the recessive model analysis involved comparing homozygous variants to the combined heterozygous and homozygous wild-type genotypes.

Statistical computations were performed using IBM SPSS Statistics version 25. Categorical variables were analyzed using the chi-square test, and the association risks were quantified as odds ratios with 95% confidence intervals. A p-value of less than 0.05 was set as the threshold for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged between 1 day and 90 days (under 3 months)
* Hospitalized for evaluation of suspected invasive bacterial infections
* Informed consent obtained from parent(s) or legal guardian(s)
* Blood, urine, cerebrospinal fluid (CSF), or stool samples collected within 72 hours of admission
* Genetic material (blood sample) available for DNA extraction

Exclusion Criteria:

* Known or suspected congenital immunodeficiency
* Previous diagnosis of genetic syndromes affecting immune function
* Major congenital anomalies or chromosomal abnormalities
* Antibiotic therapy initiated more than 24 hours before sample collection
* Parental refusal to participate or withdraw consent

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Correlation between specific gene polymorphisms and the occurrence of invasive bacterial infections in infants under 3 months | 2 weeks
  This outcome measures the correlation between the presence of the following gene polymorphisms:
  TLR4 rs2149356 (c.261-468T>G),
  LTA rs2229094 (c.37T>C), and
  RFP175 rs1585110 (c.246+8853G>A), and the occurrence of laboratory-confirmed invasive bacterial infections (IBI) in infants aged <3 months.
  Genotyping will be performed using PCR-based methods. IBIs will be categorized into one or more of the following based on predefined diagnostic criteria:
  Meningitis: confirmed by cerebrospinal fluid (CSF) pleocytosis and laboratory indicators of bacterial infection in CSF.
  Pneumonia: diagnosed based on auscultatory findings and radiographic evidence of pulmonary infiltrates.
  Sepsis and bacteremia: identified by positive blood cultures.
  Urinary tract infection: defined by a significant number of bacterial colonies in urine obtained by sterile catheterization.
  Invasive bacterial gastroenteritis: diagnosed by isolation of pathogenic bacteria in stool cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Yurtseven, MD, Principal Investigator — Ege University, School of Medicine Department of Pediatrics, Izmir, Turkey.
Locations (2):
- Turkey (Türkiye) (2):
  - Ege University School of Medicine, Izmir, İzmir
  - Ege University School of Medicine, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gomez B, Mintegi S, Bressan S, Da Dalt L, Gervaix A, Lacroix L; European Group for Validation of the Step-by-Step Approach. Validation of the "Step-by-Step" Approach in the Management of Young Febrile Infants. Pediatrics. 2016 Aug;138(2):e20154381. doi: 10.1542/peds.2015-4381. Epub 2016 Jul 5. PMID 27382134
- [Background] Carrasco-Colom J, Jordan I, Alsina L, Garcia-Garcia JJ, Cambra-Lasaosa FJ, Martin-Mateos MA, Juan M, Munoz-Almagro C. Association of Polymorphisms in IRAK1, IRAK4 and MyD88, and Severe Invasive Pneumococcal Disease. Pediatr Infect Dis J. 2015 Sep;34(9):1008-13. doi: 10.1097/INF.0000000000000779. PMID 26075815
- [Background] Ladhani SN, Davila S, Hibberd ML, Heath PT, Ramsay ME, Slack MP, Pollard AJ, Booy R. Association between single-nucleotide polymorphisms in Mal/TIRAP and interleukin-10 genes and susceptibility to invasive haemophilus influenzae serotype b infection in immunized children. Clin Infect Dis. 2010 Oct 1;51(7):761-7. doi: 10.1086/656236. PMID 20804371
- [Background] Zhao J, Gu Q, Wang L, Xu W, Chu L, Wang Y, Li Z, Wu S, Xu J, Hu Z, Shu Q, Fang X. Low-Copy Number Polymorphism in DEFA1/DEFA3 Is Associated with Susceptibility to Hospital-Acquired Infections in Critically Ill Patients. Mediators Inflamm. 2018 May 22;2018:2152650. doi: 10.1155/2018/2152650. eCollection 2018. PMID 29950924
- [Background] Chen Q, Yang Y, Hou J, Shu Q, Yin Y, Fu W, Han F, Hou T, Zeng C, Nemeth E, Linzmeier R, Ganz T, Fang X. Increased gene copy number of DEFA1/DEFA3 worsens sepsis by inducing endothelial pyroptosis. Proc Natl Acad Sci U S A. 2019 Feb 19;116(8):3161-3170. doi: 10.1073/pnas.1812947116. Epub 2019 Feb 4. PMID 30718392
- [Background] Delongui F, Carvalho Grion CM, Ehara Watanabe MA, Morimoto HK, Bonametti AM, Maeda Oda JM, Kallaur AP, Matsuo T, Reiche EM. Association of tumor necrosis factor beta genetic polymorphism and sepsis susceptibility. Exp Ther Med. 2011 Mar;2(2):349-356. doi: 10.3892/etm.2011.213. Epub 2011 Jan 20. PMID 22977509
- [Background] Esposito S, Bosis S, Orenti A, Spena S, Montinaro V, Bianchini S, Zampiero A, Principi N. Genetic polymorphisms and the development of invasive bacterial infections in children. Int J Immunopathol Pharmacol. 2016 Mar;29(1):99-104. doi: 10.1177/0394632015622961. Epub 2015 Dec 18. PMID 26684632
- [Derived] Yurtseven A, Durmusalioglu EA, Turan B, Saz EU. Correlation between single nucleotide polymorphisms in TLR4, LTA and RFP175 genes and susceptibility to invasive bacterial infections in infants under three months of age: A case control study. Pak J Med Sci. 2025 Dec;41(12):3498-3502. doi: 10.12669/pjms.41.12.12651. PMID 41450988